CLINICAL TRIAL: NCT05744531
Title: Evaluation of the Effect of Internet-based Parenting Education Based on the Information -Motivation-Behavioral Skills (IMB) Model on Maternal and Paternal Attachment
Brief Title: Internet Based Parenting Education and Information -Motivation-Behavioral Skills (IMB) Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semra TUNCAY YILMAZ (Other)
Collaborators: Semra TUNCAY YILMAZ (Unknown)
Responsible Party: Sponsor-Investigator, Semra TUNCAY YILMAZ, Principal Investigator, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: aybu sbe
Record Dates: First submitted 2022-03-22; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Parenting; Maternal-Fetal Relations; Paternal Behavior
Keywords: maternal attachment; parenteral attachment; parentering education; prenatal attachment; paternal attachmnet; internet-based education; Information-Motivation-Behavioral Skills (IMB) Model
MeSH Terms: interventions — Models, Biological

STUDY DESIGN:
Intervention Model Description: There will be two group. One is interventional group; other is control group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The volunteer and the researcher (caregiver) before agreeing to participate in the study will not know which group they will be in. After accepting the research, the participant and the researcher will know who will be in which group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education group (Experimental): The healthy pregnant women and their spouses meeting the inclusion criteria were determined by randomization according to the order of application to the antenatal clinic. A guide to providing access to internet-based education, training booklet and attachment diary was given to the pregnant women and their spouses in the education group .Internet-based Parenting education based on the Information-Motivation-Behavioral Skills (IMB) Model was given to the pregnant women and their spouses in the education group , once a week between 31 and 34 weeks of gestation, for a total of 4 times. . Internet-based counseling was given to the pregnant women and their spouses in the education group as part of the motivation step of the model,
  Interventions: Other: Internet-based Parenting Education based on the information -Motivation-Behavioral Skills (IMB) Model
- control group (No Intervention): The healthy pregnant women and their spouses meeting the inclusion criteria were determined by randomization according to the order of application to the antenatal clinic. A guide to providing access to internet-based education, training booklet and attachment diary was not given to the pregnant women and their spouses in the control group. No training was given to the pregnant women and their spouses in the control group.Counseling was not provided to the pregnant women and their spouses in the control group. .

INTERVENTIONS:
Other: Internet-based Parenting Education based on the information -Motivation-Behavioral Skills (IMB) Model — Internet-based Parenting Education based on the information -Motivation-Behavioral Skills (IMB) Model
  Arms: education group

SUMMARY:
In this study, it was aimed to evaluation of the effect of internet-based parenting education based on the information -motivation-behavioral skills (ımb) model on maternal and paternal attachment.

DETAILED DESCRIPTION:
Healthy pregnant women and their spouses participated in this study. Pregnant women and their spouses who met the research criteria were identified and randomized as intervention and control groups according to the order of application to antenatal clinic.

This study was carried out in two stages. In the first stage of the study pregnant women in both groups filled in the İndividual İnformation Form/ Mother and Prental Attachment İnventory. Spouses in both groups filled in the İndividual İnformation Form/ Father and Intrauterine Father Attachment Scale. A guide to providing access to internet-based education, training booklet and attachment diary was given to the pregnant women and their spouses in the intervention group. A guide to providing access to internet-based education, training booklet and attachment diary was not given to the pregnant women and their spouses in the control group.

In the second phase of the study; Internet-based Parenting education based on the Information-Motivation-Behavioral Skills (IMB) Model was given to the pregnant women and their spouses in the intervention group, once a week between 31 and 34 weeks of gestation, for a total of 4 times. No training was given to the pregnant women and their spouses in the control group. Prental Attachment Inventory was applied online to the pregnant women in both groups at 35th gestational week. The intrauterine Father Attachment Scale was applied online to the spouses in both groups at the 35th gestational week. Internet-based counseling was given to the pregnant women and their spouses in the intervention group as part of the motivation step of the model. This counseling was applied twice, the first between 36 and 38 weeks of gestation and the second between 20 and 40 days after delivery. Counseling was not provided to the pregnant women and their spouses in the control group. Within the scope of the behavioral skills step of the model, Maternal Attachment Inventory was applied to the mothers in the intervention group, and Paternal Infant Attachment Scale was applied to the fathers in the intervention group online at the 3nd month postpartum. The Mother Attachment Inventory was administered online to the mothers in the control group, and the Paternal Infant Attachment Scale was administered online to the fathers in the control group in the thirth month after birth.

Parameters to Look for:

In this study, it is aimed to Evaluate the Effect of Internet-based Parenting Education based on the Information-Motivation-Behavioral Skills (IMB) Model on Maternal and Paternal Attachment. Within the scope of the study, Prental Attachment İnventory scores of the pregnant women in the intervention and control groups were compared before and after the education. In addition, Maternal Attachment Inventory scores of mothers in the intervention and control groups in the postpartum period were compared. The intrauterine Father Attachment Scale scores of the fathes in the intervention and control groups were compared before and after the education. Paternal Infant Attachment Scale score in the 3nd month after birth were compared between fathers in the intervention and control groups.

Population of the Study Group:

The population of the study consisted of primiparous pregnant women and their spouses who applied to Ankara City Hospital Gynecology and Obstetrics antenatal clinic.

Sample of the Study Group: The sample of the study was calculated based on the Atalay and Saydam (2014) study results (Maternal Attachment Scale (MBI): Experimental Group X̅+SD: 101.24 ± 4.60 and Control Group X̅+SD: 96.00 9.09) (124). Analysis In Gpower version 3.1.9.7, the effect size (0.727) was calculated according to the power analysis using ''t tests-Means: Difference between two independent means (two groups) '' statistic, with α= 0.05 error level and 95% power. its size; 51 couples in the intervention group and 51 couples in the control group, a total of at least 102 couples . Since the dropout rate in the reference study was 20%, in accordance with this rate, it was planned to carry out the study with a total of 120 couples by adding a total of 18 couples, 9 couples to each group.Random Allocation Software program was used for the randomization of the groups.

Evaluation of Data: Research data will be evaluated in computer environment with appropriate statistical methods. IBM SPSS Statistics 23.0 program was used for statistical analysis and calculations. Statistical significance level was accepted as p<0.05. The conformity of the numerical variables to the normal distribution was evaluated with the Shapiro-Wilk test. The difference between the two independent groups was assessed t test and the Mann-Whitney U test . The relationship between two independent categorical variables was assessed via chi-square analysis

Data Collection Tools:

1.İndividual İnformation Form/ Mother, 2. Prental Attachment İnventory, 3. İndividual İnformation Form/ Father , 4. Intrauterine Father Attachment Scale 5. Maternal Attachment Inventory, 6. Paternal Infant Attachment Scale

ELIGIBILITY:
Inclusion Criteria:

Selection criteria for pregnant women

* Those between the ages of 18 - 35,
* At least primary school graduate,
* First pregnancy and 28 th- 30th gestational week,
* Not having a chronic health problem before pregnancy (diabetes mellitus, hypertension, kidney failure, liver failure, epilepsy, etc.),
* Those who do not have a risky pregnancy (gestational diabetes, preeclampsia, multiple pregnancy, etc.) and continue their antenatal follow-up,
* No diagnosed psychiatric problem (Anxiety, anxiety disorder, depression, bipolar etc.),
* Speaking Turkish and not having any communication barriers,
* Not a member of health sciences,
* Those who have not participated in parenting education before,
* Having a healthy spouse/partner,
* Having access to the Internet, computer and smart phone,

Selection criteria for fathers

* Those between the ages of 18 - 35,
* At least primary school graduate,
* No diagnosed psychiatric problem (Anxiety, anxiety disorder, depression, bipolar etc.),
* Speaking Turkish and not having any communication barriers,
* Not a member of health sciences,
* Those who have not participated in parenting education before,
* Having a healthy spouse/partner,
* Having access to the Internet, computer and smart phone,

Exclusion Criteria:

* Inclusion of the mother in the risky pregnancies group (bleeding, preeclampsia, premature birth, etc.),
* Taking the newborn to the intensive care unit,
* Incomplete filling of data collection forms,
* If one or any of the parents has stopped participating in the study; both individuals will be excluded from the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Maternal Attachment | 3nd month after birth
  maternal attachment level measured by Maternal Attachment Inventory .It is a 4-point Likert-type scale with 26 items. Each item directly. It is always (a) = 4 points, often (b) = 3 points, sometimes (c) = 2 points, and never (d) = 1 point.Test scored between 26-104. A high score indicates high maternal attachment
Paternal Infant Attachment Scale | 3nd month after birth
  paternal attachment level measured by Paternal Infant Attachment Scale. The scale has three sub-dimensions and 19 items. The sub-dimensions of the scale include "Patience and Tolerance", "Pleasure in Interaction", "Love and Pride". Each item of the scale is scored between one and five points, and the score that can be obtained from the scale varies between 19 and 95.

SECONDARY OUTCOMES:
Prenatal Attachment | within 1 week after education
  Prenatal attachment level measured by Prental Attachment İnventory. The scale is applied in the prenatal period from the 28th gestational week until the birth. The PCI consists of 21 items in total and the items in the scale are scored on a four-point Likert scale that can range from 1 to 4. A minimum of 21 and a maximum of 84 points can be obtained from the scale.
  Test scored between 21-84
Intrauterine Father Attachment Scale | within 1 week after education
  Intrauterine Father Attachment level measured by Intrauterine Father Attachment Scale . The scale consists of 23 items and is a four-point Likert scale. The scale does not have a cutoff point. The higher the mean score obtained from the scale, the higher the level of attachment of fathers to their babies Test scored between 23-92.

CONTACTS AND LOCATIONS:
Overall Officials: özlem Moraloğlu Tekin, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manav AI, Gozuyesil E, Tar E. The Effects of the Parenting Education Performed through Whatsapp on the Level of Maternal-Paternal and Infant Attachment in Turkey. J Pediatr Nurs. 2021 Nov-Dec;61:e57-e64. doi: 10.1016/j.pedn.2021.04.018. Epub 2021 Apr 26. PMID 33926747

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT05744531/Prot_SAP_ICF_000.pdf